CLINICAL TRIAL: NCT02801435
Title: A Single-Center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Icotinib Hydrochloride Cream in Patients With Mild to Moderate Psoriasis
Brief Title: Icotinib Hydrochloride Cream in Patients With Mild to Moderate Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BD-ICC-I01
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Psoriasis
Keywords: EGFR inhibitor; topical agent; psoriasis; phase 1
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1-Experimental (Experimental): 8 patients with mild to moderate psoriasis will be randomized to receive 0.5% Icotinib hydrochloride cream, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: 0.5% Icotinib hydrochloride cream
- Cohort 1-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Placebo
- Cohort 2-Experimental (Experimental): 8 patients with mild to moderate psoriasis will be randomized to receive 1.0% Icotinib hydrochloride cream, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: 1.0% Icotinib hydrochloride cream
- Cohort 2-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Placebo
- Cohort 3-Experimental (Experimental): 8 patients with mild to moderate psoriasis will be randomized to receive 2.0% Icotinib hydrochloride cream, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: 2.0% Icotinib hydrochloride cream
- Cohort 3-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Placebo
- Cohort 4-Experimental (Experimental): 8 patients with mild to moderate psoriasis will be randomized to receive 4.0% Icotinib hydrochloride cream, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: 4.0% Icotinib hydrochloride cream
- Cohort 4-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 4 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.5% Icotinib hydrochloride cream — Topical administration for twice daily
  Other Names: no other name
  Arms: Cohort 1-Experimental
Drug: 1.0% Icotinib hydrochloride cream — Topical administration for twice daily
  Other Names: no other name
  Arms: Cohort 2-Experimental
Drug: 2.0% Icotinib hydrochloride cream — Topical administration for twice daily
  Other Names: no other name
  Arms: Cohort 3-Experimental
Drug: 4.0% Icotinib hydrochloride cream — Topical administration for twice daily
  Other Names: no other name
  Arms: Cohort 4-Experimental
Drug: Placebo — Topical administration for twice daily
  Other Names: Blank cream
  Arms: Cohort 1-Placebo; Cohort 2-Placebo; Cohort 3-Placebo; Cohort 4-Placebo

SUMMARY:
This is a phase I study to evaluate the safety, tolerability and pharmacokinetics of Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis.

DETAILED DESCRIPTION:
Icotinib Hydrochloride is a small-molecule epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor, which has been approved for the treatment of advanced nonsmall- cell lung cancer (NSCLC) in China in its oral form. As EGFR is implicated in the pathogenesis of psoriasis, icotinib hydrochloride is being developed as a cream for the treatment of mild to moderate psoriasis. This is a single-center, randomized, doubleblind, placebo-controlled study of 0.5%, 1.0%, 2.0%, 4.0% icotinib hydrochloride cream by topical administration. Icotinib hydrochloride cream will be applied to subjects with mild to moderate psoriasis. Approximately 40 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis for at least six months with multiple treatable area (i.e. the lesion should not only on the face, scalp, genitals or skinfolds) of plaque psoriasis covering less than 10% of the total Body Surface Area (BSA), affected area on the limb and/or trunk≥ 1% BSA. A Target Plaque Area (TPA)≥9 cm2, with a Target Plaque Severity Score(TPSS)≥ 5, and induration subscore≥2.
* Male participants should be ≥ 50 kg, female participants should be ≥ 45 kg; BMI should be between 19 and 28 kg/m2 (inclusive)
* In good health, with no history of diseases of major organs and no abnormality found on physical examination and vital signs
* Non-allergic, with no known history of drug allergy
* Men and women of childbearing potential must agree to use a contraceptive regimen agreed by the doctor during the trial. Female subjects that are on hormonal contraceptives must continue using the same hormonal contraceptive as that was used in the past 3 months, with the same route of administration and the same dose during the study
* Have signed a written informed consent before entering the study

Exclusion Criteria:

* Psoriasis guttata, psoriasis punctata, erythrodermic psoriasis, pustular psoriasis, psoriasis arthritis
* Any dermatological disease that might interfere psoriasis clinical evaluation or bring the subject in danger, or have other serious dermatological disease other than psoriasis.
* Have received underlying treatments before entering the trial:

Topical anti-psoriasis treatment in 2 weeks, e.g. corticosteroids, retinoids acid, anthranol, tars, keratolytics. Vitamin D analogues or local immune regulator treatment in 4 weeks; Emollient or cosmetics in 24 hours; Any psoriasis vaccine, or have participated in any psoriasis vaccine trial; Biologics treatment in 12 weeks, e.g. Alefacept, Etanercept, Infliximab, Adalimumab, Ustekinumab, Efalizumab; Any phototherapy or systemic treatment in 4 weeks, e.g. corticosteroids, methotrexate, retinoids acids, ciclosporin; Long time exposure to natural light or artificial UV, or will have such exposure; Use of drug known to harm certain organ in 12 weeks; Participated in any clinical trial in 4 weeks, or have plan to participate any trial during treatment period;

* Any clinically significant central nervous, cardiac, hepatic, renal, gastrointestinal, respiratory, metabolic or musculoskeletal system disease history, or other pathological/physiological condition that might disrupt the trial result
* Alanine transaminase(ALT), aspartate aminotransferase (AST), total bilirubin>1.5 Upper Limit Normal (ULN), creatinine>ULN
* History of postural hypotension, or allergic diseases (asthma, urticaria, atopic dermatitis or rhinitis)
* Pulmonary disease demonstrated by chest X-ray examination
* Physically or mentally disabled
* Positive for Hepatitis B Surface Antigen (HBsAg), hepatitis C or anti-HIV test
* Know allergic to active ingredient or excipient of the investigational product
* Excessive smoker(>10 cigarettes per day), or excessive alcohol intake (>15g absolute alcohol per day, equal to 450ml beer, 150ml wine or 50ml low-alcohol Chinese liquor)
* Excessive drinking of tea, coffee or caffein-containing beverage (>8 glasses per day)
* Drug abuser
* Poor compliance
* Under gestation or lactation period
* Other subject that in the investigator's opinion unsuitable to be enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09-17 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Safety in patients with mild to moderate psoriasis | 28 days
  Incidence and severity of Adverse Events (AE), Physical Examinations, Vital signs (temperature, Heart Rate (HR), BP and respiration); Clinical laboratory assessments (serum chemistry, hematology, C-reactive protein , fecal and urinalysis); ECG;

SECONDARY OUTCOMES:
Tolerance-related skin reactions in patients with mild to moderate psoriasis at the treatment site | 28 days
  Skin irritation and allergy observation (including redness, swelling,rash, itching, pain) recorded by grades

OTHER OUTCOMES:
Lesion severity | 28 days
  Erythema , scale , thickness of target site on patients with mild to moderate psoriasis
Lesion area | 28 days
Psoriasis Area and Severity Index (PASI) Scores in patients with mild to moderate psoriasis | 28 days
Physician's Global Assessment(PGA) in patients with mild to moderate psoriasis | 28 days
Dermatology Life Quality Index (DLQI) in patients with mild to moderate psoriasis | 28 days
Time maximum concentration observed(tmax) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 12 hours
Peak plasma concentration (Cmax) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 12 hours
Area under the plasma concentration versus time curve(AUC) of single-dose Icotinib Hydrochloride Cream from zero(0) hours to time (t) in patients with mild to moderate psoriasis | 12 hours
Area under the plasma concentration versus time curve(AUC) of single-dose Icotinib Hydrochloride Cream from zero (0) hours to infinity (∞) in patients with mild to moderate psoriasis | 12 hours
Half life(t1/2) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 12 hours
Time maximum concentration observed(tmax) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 24 hours
Stable peak plasma concentration (Cmaxss) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 24 hours
Area under the plasma concentration versus time curve(AUC) of repeat-dose Icotinib Hydrochloride Cream from zero(0) hours to time (t) in patients with mild to moderate psoriasis | 24 hours
Area under the plasma concentration versus time curve(AUC) of repeat-dose Icotinib Hydrochloride Cream from zero (0) hours to infinity (∞) in patients with mild to moderate psoriasis | 24 hours
Half life(t1/2) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, Principal Investigator — The Second Affiliated Hospital of Zhejiang University School of Medicine (SAHZU); Zourong Ruan, Principal Investigator — The Second Affiliated Hospital of Zhejiang University School of Medicine (SAHZU)
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No